CLINICAL TRIAL: NCT04635020
Title: A Prospective Randomised Trial Comparing Selective Laser Trabeculoplasty (SLT) and iStent Trabecular Micro-bypass Stent Implantation Combined With Cataract Surgery in Exfoliation Glaucoma
Brief Title: Comparison Of iStent to Laser in Exfoliation Glaucoma Helsinki Study Group
Acronym: COILEH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Prof. Mika Harju, MD, professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123123
Record Dates: First submitted 2020-10-29; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Exfoliation Glaucoma; Cataract
Keywords: SLT; iStent
MeSH Terms: conditions — Exfoliation Syndrome; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Stable glaucoma iStent (Experimental): Cataract surgery combined with iStent inject
  Interventions: Procedure: iStent; Procedure: Cataract surgery
- Stable glaucoma SLT-laser (Experimental): Cataract surgery combined with SLT-laser 1 month after surgery
  Interventions: Procedure: SLT-laser; Procedure: Cataract surgery
- Stable glaucoma (Active Comparator): Cataract surgery
  Interventions: Procedure: Cataract surgery
- Unstable glaucoma iStent (Experimental): Cataract surgery combined with iStent inject
  Interventions: Procedure: iStent; Procedure: Cataract surgery
- Unstable glaucoma SLT-laser (Experimental): Cataract surgery combined with SLT-laser 1 month after surgery
  Interventions: Procedure: SLT-laser; Procedure: Cataract surgery

INTERVENTIONS:
Procedure: iStent — 2 trabecular Stent injected at the end of the cataract surgery to the trabecular meshwork
  Other Names: Trabecular Micro-Bypass Stent System Model G2-M-IS, Glaukos Corporation, San Clemente, California
  Arms: Stable glaucoma iStent; Unstable glaucoma iStent
Procedure: SLT-laser — 1 month after cataract surgery laser treatment to the trabecular meshwork (100 applications, 360 degrees)
  Other Names: Selective laser trabeculoplasty
  Arms: Stable glaucoma SLT-laser; Unstable glaucoma SLT-laser
Procedure: Cataract surgery — Conventional cataract surgery

SUMMARY:
The purpose of the study is to investigate the efficacy of an iStent trabecular microbypass stent compared to selective laser trabeculoplasty in combination with cataract surgery in eyes with exfoliation glaucoma (EXF)

DETAILED DESCRIPTION:
Exfoliation glaucoma patients with significant cataracts are being informed about the study and potential risks, all patients giving written informed consent will undergo screening to determine eligibility for study entry. Patient´s glaucoma is classified into stable or unstable glaucoma groups with their current glaucoma medication. Patients meeting the eligibility requirements of stable glaucoma will be randomised to cataract surgery combined with iStent (65 patients), II SLT (65 patients) or III cataract surgery alone (25 patients) and patient with unstable glaucoma will be randomised to cataract surgery combined with I iStent (65 patients), II SLT (65 patients).

ELIGIBILITY:
Inclusion Criteria:

* Signed consent of information
* Clinical significant cataract
* Able to attend 12 month period
* Mild to moderate exfoliation glaucoma according to European glaucoma society guidelines (EGS)
* Group I stable glaucoma (IOP within individual target IOP), and group II unstable glaucoma (IOP above individual target IOP) with baseline glaucoma medication
* Target IOP ≥16
* Able to understand Finnish, Swedish or English

Exclusion Criteria:

* Clinical set target IOP < 16 mmHg in advanced glaucoma
* Baseline IOP prior to enrolment ≥30 mmHg, and ≥3 glaucoma medications
* Closed angle
* Congenital angle anomaly
* Clinically significant corneal dystrophy or other hindering corneal condition
* Unable to use topical medical therapy
* Central corneal thickness of less than 480um or more than 620um
* Active uveitis, cystic macular edema (CME), exudative age-related macular degeneration, proliferative diabetic retinopathy or clinical significant macular edema, intraocular neoplasm, intraocular injections, intraocular lens luxation, phacodonesis.
* Previous intraocular surgery, refractive surgery or cycloablation
* Two or more prior SLT or laser trabeculoplasty
* Unable to participate due to another medical disease or condition
* Participating in another clinical trial

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Group I: Change in the number of IOP lowering medications compared to baseline | 12 months
  Accountability of IOP lowering medications used by the patient
Group II: Change in the IOP compared to baseline | 12 months
  IOP measured by Goldmann aplanation tonometry (GAT)

SECONDARY OUTCOMES:
Group I: Change in the IOP compared to baseline | 12 months
  IOP measured by GAT
Group II: Change in the number of IOP lowering medications compared to baseline | 12 months
  Accountability of IOP lowering medications used by the patient

OTHER OUTCOMES:
Group I and II: Number of patients with secondary glaucoma surgery | 10 years
  Number of patients with secondary glaucoma surgery at 10 years from baseline is counted

CONTACTS AND LOCATIONS:
Overall Officials: Mika Harju, MD, prof., Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No